CLINICAL TRIAL: NCT05320913
Title: Pericapsular Nerve Group (PENG) Block Combined With Periarticular Multimodal Drug Injection (PMDI) Versus Isolated PMDI for Pain Management After Total Hip Arthroplasty: a Randomized Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 4-2021-1482
Record Dates: First submitted 2022-04-03; First posted 2022-04-11 (Actual); Last update posted 2022-05-03 (Actual); Status verified 2022-05

CONDITIONS: Total Hip Arthroplasty, Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pericapsular nerve group(PENG) block combined with periarticular multimodal drug injection (PMDI) (Experimental): Participants receiving pericapsular nerve group(PENG) block combined with periarticular multimodal drug injection (PMDI)
  Interventions: Procedure: Pericapsular nerve group(PENG) block combined with periarticular multimodal drug injection (PMDI)
- isolated periarticular multimodal drug injection (PMDI) (Active Comparator): Arm Description: Participants receiving isolated periarticular multimodal drug injection (PMDI)
  Interventions: Procedure: isolated periarticular multimodal drug injection (PMDI)

INTERVENTIONS:
Procedure: Pericapsular nerve group(PENG) block combined with periarticular multimodal drug injection (PMDI) — periarticular local anesthetic infiltration with 120 mg of ropivacaine, epinephrine 0.2 mg and 30 mg of ketorolac diluted with normal saline to a total volume of 40 mL. + PENG block with ropivacaine 40 mg and epinephrine 0.1 mg with normal saline to a total volume of 20 mL
  Other Names: PENG + PMDI block
  Arms: Pericapsular nerve group(PENG) block combined with periarticular multimodal drug injection (PMDI)
Procedure: isolated periarticular multimodal drug injection (PMDI) — periarticular local anesthetic infiltration with 150 mg of ropivacaine, epinephrine 0.3 mg and 30 mg of ketorolac diluted with normal saline to a total volume of 50 mL
  Other Names: Isolated PMDI block
  Arms: isolated periarticular multimodal drug injection (PMDI)

SUMMARY:
Adequate pain control after total hip arthroplasty is crucial for early ambulation and patient satisfaction. However, there is no consensus about optimal pain control after post operation. In general, the periarticular multimodal durg injection block has been done for pain control in primary total hip arthroplasty. The pericapsular nerve group (PENG) block has been recently introduced a new technique for blockade of the articular branches of the femoral, obturator and accessory obturator nerves. PENG block is possible to provide sufficient analgesia and preserve lower limb muscle strength. The investigators will compare PENG and PMDI block with isolated PMDI block in patients undergoing total hip arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 19 years old or older, with American Society of Anesthesiologists Physical Status 1-3, and scheduled for elective unilateral total hip arthroplasty

Exclusion Criteria:

1. Allergy or intolerance to any of the drugs used in the study
2. Hepatic or renal insufficiency
3. Opioid dependency
4. Coagulopathy
5. Pre-existing neurologic or anatomic deficits in the lower extremities
6. Severe psychiatric illness

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2022-04-04 (Actual); Primary Completion 2023-12-13 (Estimated); Study Completion 2023-12-13 (Estimated)

PRIMARY OUTCOMES:
Numeric rating scale pain score | at 24 hours postoperatively
  Pain intensity at rest evaluated by an 11-point numeric rating scale (NRS: 0 = no pain, 10 = worst imaginable pain) at 24 hours postoperatively

SECONDARY OUTCOMES:
Pain score measured at 6 hours postoperatively and 48 hours postoperatively | Pain score measured at 6 hours postoperatively and 48 hours postoperatively
  Pain intensity at rest evaluated by an 11-point numeric rating scale (NRS: 0 = no pain, 10 = worst imaginable pain) at 6 hours postoperatively and 48h postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Kwankyu Park, Principal Investigator — Department of orthopaedic surgery, Yonsei University College of Medicine
Locations (1):
- Yonsei University Health System, Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Cho HS, Lee BR, Kwon HM, Park JY, Ham HW, Lee WS, Park KK, Lee TS, Choi YS. Pericapsular Nerve Group Block with Periarticular Injection for Pain Management after Total Hip Arthroplasty: A Randomized Controlled Trial. Yonsei Med J. 2025 Apr;66(4):233-239. doi: 10.3349/ymj.2024.0098. PMID 40134083